CLINICAL TRIAL: NCT02162979
Title: A Double-Blind, Placebo-Controlled, Cross-Over Study of Sildenafil (Viagra) for the Treatment of Dyskinesias in Parkinson's Disease
Brief Title: Sildenafil (Viagra) for the Treatment of Dyskinesias in Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough subjects.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 52031
Record Dates: First submitted 2007-12-26; First posted 2014-06-13 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; dyskinesia; treatment; motor complications
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Viagra (Experimental): subjects will be randomized to active treatment for 2 weeks, washout for 1 week, then enter the other study arm for two weeks.
  Interventions: Drug: sildenafil
- Placebo comparator (Placebo Comparator): subjects will be randomized to placebo treatment for 2 weeks, washout for 1 week, then enter the other study arm for two weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 50mg BID for 2 weeks
  Other Names: Viagra
  Arms: Viagra
Drug: Placebo
  Arms: Placebo comparator

SUMMARY:
This study is to determine if Viagra is effective in reducing dyskinesias in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease.
2. Age > 40 years.
3. willingness and ability to comply with the study requirements and give informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease, Hoehn and Yahr stage 2.0 to 4.0.
2. Presence of drug-induced dyskinesias
3. Age>40 years.
4. Willingness and ability to comply with the study requirements and give informed consent.

Exclusion Criteria:

1. Atypical parkinsonian syndrome due to drugs, metabolic disorders, encephalitis, or degenerative diseases.
2. History of stereotaxic brain surgery.
3. Clinical history of dementia.
4. Known major psychiatric disorder, major depression, schizophrenia. Known alcoholism or substance dependence within previous 12 months.
5. History of major hematological, renal, or hepatic abnormalities.
6. Known coronary artery disease including angina or myocardial infarction within the last 6 months. Significant cardiovascular disease including cardiac failure, unstable angina or life-threatening arrhythmia within the last 6 months.
7. History of stroke within the last 6 months.
8. Abnormal EKG consistent with cardiac ischemia.
9. Treatment with nitrates. Nitrates or any NO donors in any dosage form (oral, sublingual, transdermal, inhalation, or aerosols).
10. Malignant hypertension or SBP . 180 or <90, or DBP .110 or <50.
11. History of priapism.
12. Known history of retinitis pigmentosa.
13. Positive pregnancy test.
14. History of bleeding disorder.
15. Patients with active peptic ulcer disease associated with bleeding.
16. Unwillingness to use adequate contraceptive methods if of childbearing potential.
17. Patients with medical or psychological condition or social circumstances that would impair their ability to participate in the study.
18. Use of Viagra or any experimental drugs within 30 days of screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Swope, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Documentation regarding the randomization of the two enrolled participants cannot be located. Therefore no meaningful data are available for entry in the data tables.
Groups:
- Placebo Comparator: subjects will be randomized to placebo treatment for 2 weeks, washout for 1 week, then enter the other study arm for two weeks.
  Placebo
Period: Overall Study
Arm/Group | Viagra | Placebo Comparator
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Viagra | Placebo Comparator | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Change in Duration of Dyskinesia.
Time Frame: 2 weeks
Arm/Group | Viagra | Placebo Comparator
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change in "on" Time
Description: "on" time is the period in which the subject is symptom free. We will track the amount of time the subject is considered symptom free before and after treatment. This value will be represented as a percent change.
Time Frame: 4 weeks
Arm/Group | Viagra | Placebo Comparator
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Dose of Anti-parkinsonian Medications
Time Frame: 7 weeks
Arm/Group | Viagra | Placebo Comparator
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Viagra | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes